CLINICAL TRIAL: NCT06458114
Title: Feeling of Caregivers After a Palliative Management in Delivery Room of Extreme Premature Babies Not Eligible for Intensive Care : a French Qualitative and Quantitative Monocentric Study.
Brief Title: Feeling of Caregivers After a Palliative Management of Extreme Premature Babies in Delivery Room.
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO22027
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Caregiver Feeling
Keywords: Caregiver feeling; Palliative care; Delivery room; Extremely preterm birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of caregiver feeling — The study group includes any caregiver who supported an extremely preterm newborn in a palliative care approach in the delivery room with as intervention type a questionnaire and individual semi-structured interview.

SUMMARY:
Introduction :

The birth of a child is usually a happy event that caregivers working in delivery rooms share with families.

Unfortunately, newborns sometimes need palliative care as soon as birth occurs.

In France, neonates who were liveborn under 24+0 weeks amenorrhea (date of last mentrual period) or weighing less than 500 grams) usually have non resuscitation in delivery room [Ancel 2020]. Some of them are considered as viable (referring to World Health Organisation definition : either term ≥ 22 + 0 amenorrhea week or birth weight ≥ 500 grams), others as nonviable (term < 22 AW and birth weight ≤500 grams).

In France, legislative development over last two decades have allowed the emergence of palliative care in delivery room. In a French survey in 2016, 83% of maternities were confronted at least once a year with this situation.

DETAILED DESCRIPTION:
In France as in other countries, published studies concerning palliative care for extremely premature babies focused on the " grey zon " period, but not on the nonviable preterm infants (also called late miscarriage) who have signs of life at birth. Only a fairly recent French book of 735 pages exclusively dedicated to the palliative approach in perinatal medicine, reports in a single chapter the existence of palliative care in extremely non-viable premature newborns.

There is a paucity of articles about the actual experience of caregivers confronted to palliative care of extremely preterm babies, viable or non viable, primarily studies in the so-called "gray" literature. Thus, a midwifery graduation thesis describes the experience of midwives in a French university hospital following the care of babies born alive between 18 and 24 weeks old . Two recent reviews explore the notion of resilience of caregivers who have been involved in perinatal palliative care . A nursing graduation dissertation explores the emotions of caregivers faced with perinatal bereavement .

Primary objective: the primary objective of this both qualitative and quantitative monocentric study is to explore the feelings of caregivers (doctors, midwifes, nurse's aids, pediatric nurses) within 2 months of a palliative situation for an extremely preterm baby in a delivery room, viable or not, and not eligible for resuscitation.

Secondary objective: the secondary objective of the study is to quantify the impact of this stressful event:

* Within the first month (acute stress).
* 2 months after the event (post-traumatic stress).

Expected impact of the study:

* These care situations are not described in the scientific literature and little described in the so-called grey literature: this study aims to make them readable.
* The caregiver's feelings and the mechanisms that underlie them may differ, depending on the type of profession and links within a team: this study aims to better characterize and understand them.
* As a result, the investigators hope this study will identify avenues for work and action to better support caregivers and prevent work-related burnout.

ELIGIBILITY:
Inclusion Criteria:

* Any caregiver working at the Universitary Hospital of Reims (France) (pediatrician, obstetrician, midwife, midwife, nurse's aide, pediatric nurse, midwife student, peidatrician student).
* who cared for an extremely preterm newborn in a delivery room, with a palliative approach,
* and gave his/her consent.
* The baby must have shown at least minimal signs of vitality (that is : heartbeats, cry, respiratory movements, painful facies, gasps).
* The caregiver must has been physically present with either the newbor, or the mother, or both.

Exclusion Criteria : none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study group includes any caregiver who supported an extremely preterm newborn in a palliative care approach in the delivery room. Caregivers can be : senior pediatricians, senior obstetricians, midwifes, nurse's aides, pediatric nurses, pediatrician student, midwife student.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-07 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of caregiver feeling | 1 month
  Semi-directional interviews will be carried out with the identification of the main themes during the verbatim transcription (qualitative study).

SECONDARY OUTCOMES:
Assessment of stress | 1 month
  Revised Impact of Event Scale (IES-R) [Weiss, Brunet] scale
Assessment of stress | 2 months
  Revised Impact of Event Scale (IES-R) [Weiss, Brunet] scale

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France